CLINICAL TRIAL: NCT07039279
Title: Establishment of Hong Kong Diabesity Register and a 3-year Randomized Clinical Trial for the Investigation of the Effectiveness of a Multicomponent Integrated Care Program in Chinese With Diabesity
Brief Title: Hong Kong Diabesity Register & 3-Year Trial on Integrated Care for Chinese With Diabesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alice Pik Shan KONG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE 2025.324
Record Dates: First submitted 2025-06-04; First posted 2025-06-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Diabesity
MeSH Terms: conditions — Diabesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multicomponent Integrated Care Program (Experimental): The multicomponent integrated care program is supported by a team of endocrinologist, dietitian, psychologist and research assistant with elements including medical therapy, cognitive behavioural therapy, e-care (TourHeart + platform), artificial intelligence chatbot, biofeedback, peer support.
  Interventions: Behavioral: Multicomponent Integrated Care Program; Other: TourHeart + platform
- Control (Usual Care) (Other): Control
  Interventions: Other: TourHeart + platform

INTERVENTIONS:
Behavioral: Multicomponent Integrated Care Program — The multicomponent integrated care program is supported by a team of endocrinologist, dietitian, psychologist and research assistant with elements including medical therapy, cognitive behavioural therapy, e-care (TourHeart + platform), artificial intelligence chatbot, biofeedback, peer support
  Arms: Multicomponent Integrated Care Program
Other: TourHeart + platform — TourHeart+ is a web-based program that provides mental health services that integrate both online and offline elements, opening up new possibilities for mental well-being. Participants will be introduced to the platform but the control group will not receive follow-up action. The platform is part of the multi-intervention care program and the participants in the intervention will receive follow-up action to engage their usage of the platform.

SUMMARY:
People with diabetes and obesity (diabesity) are difficult to treat with many unmet needs requiring personalized treatment regimens, intensive counselling and emotional support. Here, we propose to conduct a pragmatic trial including 2 parts: (1) establishment of a register for Hong Kong Chinese with diabesity and through this register, identify participants consecutively to enter (2) a 3-year randomized clinical trial to assess the effects of multicomponent integrated care program supported by a team of endocrinologist, dietitian, psychologist and research assistant with elements including medical therapy, cognitive behavioural therapy, e-care, artificial intelligence chatbot, biofeedback, peer support to improve the physical and mental health in people with diabesity, with weight reduction as primary outcome. Other outcomes include cardiometabolic risk factors, diabetes distress, lifestyles and sleep hygiene.

DETAILED DESCRIPTION:
Diabetes is both a public and personal health disaster if not diagnosed, treated or managed properly. Over 60% of all cause deaths and disabilities including stroke, leg amputation, heart disease, cancer, kidney disease, depression to name but a few are causally linked to diabetes. In the United Kingdom Prospective Diabetes Study (UKPDS), a landmark clinical trial of patients with type 2 diabetes, 0.9% reduction in glycated hemoglobin (HbA1c) reduced diabetes-related microvascular complications by 12-25%. In the 10-year post-trial follow-up period, the benefits of attaining glycemic control early had a legacy effect in reducing all clinical outcomes including cardiovascular complications and death. Nonetheless, it is a worldwide phenomenon that majority of people with type 2 diabetes are not reaching glycemic goals due to clinical inertia with delayed escalation of therapy, poor treatment compliance and/or insufficient self management.

Since 1995, as part of a quality improvement program, patients attending our twice-weekly diabetic complication screening sessions at the Prince of Wales Hospital (PWH) underwent detailed documentations of clinical and biochemical information which formed the basis of the Hong Kong Diabetes Register. Data from this prospective cohorts and others have shown that obese people with type 2 diabetes are particularly difficult to treat with extremely high risk for future events. Weight control is a major therapeutic challenge which often requires cognitive-psychological-behavioral therapy (CBT) in addition to pharmacological which at times might call for surgical interventions. Many traditionally used glucose lowering agents, such as sulphonylurea and insulin, can cause weight gain, thus setting up a vicious cycle with increasing insulin resistance due to increasing levels of free fatty acids from adipose tissues. During a 6-month study, patients with type 2 diabetes treated with intensive insulin therapy dropped their HbA1c by 2.6% but gained an average of 8.7kg. Similarly, data from the UKPDS which recruited newly diagnosed type 2 diabetes, showed that patients had significant weight gain during a 10-year follow up period, particularly those on insulin therapy.

In a prospective analysis, insulin-treated type 2 diabetic patients with residual beta cell function as evidenced by high fasting serum C-peptide levels, had the highest rate of cardiovascular events of over 10%. This high event rate might be due to long disease duration, renal impairment and autonomic neuropathy with incresaed risk of hypoglycemia which substantially increased the risk of cardivoascular disease. People with diabesity have many unmet needs which require individualized therapy, intensive counselling and emotional support which cannot be adequately addressed in a busy clinic setting with 10-15 minute consultation. Besides, many patients with diabetes of working age tend to default due to competing priorities and silent nature of the disease and regrettably only to present with preventable complications after a few years.

In a series of randomized studies and disease management programs which has demonstrated the benefits of team approach, case management, quality improvement and patient empowerment on risk factor control, we have confirmed the marked benefits of using a interdisciplinary team to deliver protocol-driven care on clinical outcomes. Important features of this program included continuation of care through periodic reminders, decision support, empowerment, peer support and feedback. In a multicentre randomized study involving over 600 type 2 diabetic patients, we have demonstrated the benefits of a web-based disease management program,Joint Asia Diabetes Evaluation (JADE) program, which provides integrated and visual information to communicate personalized risks and treatment targets on reducing multiple risk factors, reducing treatment non-compliance, improving psychological health and enhancing self efficiacy in 20-30% of participants . Amongst those with negative emotions who accounted for 20% of the cohort, peer support further improved compliance and reduced hospitalization rates.

Against this background, we propose to conduct a study with 2 parts: 1) First, the establishment of Diabesity Register of Hong Kong Chinese, and through this Diabesity Register, identify eligible participants to enter: 2) a 3-year Randomized Clinical Trial (RCT) to evaluate the effectiveness of multicomponent integrated care (MIC) program in these people with diabesity.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes;
2. Obesity reaching action level as defined as body mass index (BMI) ³27.5 kg/m2 and/or waist circumference (WC) ³80cm in women and ³90cm in men;
3. Age between 18 and 50 years;
4. Able to conversate with smartphone technology and web-based program.
5. Able to read Chinese and communicate using Chinese.

Exclusion Criteria:

1. Type 1 diabetes;
2. Active malignant disease including those with history of malignant disease less than 5 years of disease-free duration;
3. Life expectancy less than 12 months;
4. Any medical illness or condition as judged by the investigators as ineligible to participate the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5% body weight reduction from baseline at year 1 | 12 months

SECONDARY OUTCOMES:
10% body weight reduction from baseline at year 1 | 12 months

OTHER OUTCOMES:
Changes in body weight | 24 months and 36 months
Blood pressure | 12 months, 24 months and 36 months
Lipid profile | 12 months, 24 months and 36 month
  Including total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, triglyceride.
Dietary energy intake | 12 months, 24 months and 36 months
  Measure by 3-days food diary.
Physical activity level | 12 months, 24 months and 36 months
  Measure by international physical activity questionnaire.
Mental health | 12 months, 24 months and 36 months
  Measure depression using Patient Health Questionnaire 9 items.
Diabetes related distress | 12 months, 24 months and 36 months
  Measure by Diabetes Distress Scale. It is a 15 item scale scoring from 1 to 6 for each questions. A higher score indicates a greater level of distress related to managing diabetes.
Health related quality of life | 12 months, 24 months and 36 months
  Measure by EuroQol Group EQ-5D questionnaire.
Presenteeism and productivity loss | 12 months, 24 months and 36 months
  Measure by Work Productivity and Activity Impairment Questionnaire: General Health.
Insomnia and its severity | 12 months, 24 months, 36 months
  Measure by Insomnia Severity Index.
Drug adherence and self-care behavior self report form | 12 months, 24 months and 36 months
  Participants will report their self care during the Joint Asia Diabetes Evaluation assessment. The following up be self-reported:
  Self-monitoring type (Self-monitoring of blood glucose/Continuous glucose monitoring/Both self-monitoring of blood glucose and continuous glucose monitoring/Urine/None) Self-monitoring in last 3 months (<once monthly/At least once monthly/At least once weekly/At least daily) Physical activity in last 3 months (No regular activity/<3 times per week/3-4 times per week/5 times per week/>5 times per week) Physical activity of moderate intensity per week (None/<150 minutes/>150 minutes) Adherence to balanced diet in last 3 months (Yes/No/Occasionally/Never) Did you ever forget to take/self-adjust diabetes mellitus drugs? (Yes/No) 0-100, rate your drug adherence level 0-100, rate your today's health status 0-100, rate your today's happiness level
Changes in the number of complications | 36 months
  Compare between 2 groups with patients in the Diabesity Register not participating in the trial as the background population.
Blood pressure | 36 months
  Compare between 2 groups with patients in the Diabesity Register not participating in the trial as the background population.
Lipid profile | 36 months.
  Compare between 2 groups with patients in the Diabesity Register not participating in the trial as the background population. Including total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, and triglyceride
Engagement with "TourHeart +" web-based program measure by modules completed by participants and frequencies of exercise completed by patients. | 12 months, 24 months and 36 months
  TourHeart+ is a web-based program that provides mental health services that integrate both online and offline elements, opening up new possibilities for mental well-being.The completion of modules and the frequency of exercise completed will be measured from backend data.
Sleep onset latency | 12 months, 24 months and 36 months
  Measure by actigraphy.
Wake after sleep onset | 12 months, 24 months and 36 months
  Measure by actigraphy.
Sleep efficiency | 12 months, 24 months and 36 months
  Measure by actigraphy.
Total sleep time | 12 months, 24 months and 36 months
  Measure by actigraphy.
Time in range | 36 months
  The duration of time of blood glucose level that is within the target glucose range (3.9-10.0 mmol/L) measure by continuous glucose monitoring.
Time above range | 36 months
  The duration of time of blood glucose level that is higher than the target range (level 1: >10.0-13.9 mmol/L, and level 2: >13.9mmol/L) measure by continuous glucose monitoring.
Time below range | 36 months
  The duration of time of blood glucose level that is below the target range (level 1: 3.0-3.8 mmol/L, and level 2: <3.0 mmol/L) measure by continuous glucose monitoring.
Glycemic variability | 36 months
  Co-efficient of variation (%CV) and mean amplitude of glycemic excursions derived from continuous glucose monitoring data.
Mean glucose | 36 months
  Measure by continuous glucose monitoring
Glucose management indicator | 36 months
  The HbA1c estimate by continuous glucose monitoring.
Percentage to achieve time in range | 36 months
  The percentage of time a person with diabetes spends within the target glucose range (3.9-10.0 mmol/L) measure by continuous glucose monitoring.
Health and disability level | 12 months, 24 months and 36 months
  Measure by the World Health Organization Disability Assessment Schedule 2.0 12-item (WHO-DAS 2.0-12item), scoring from 0-100 and a higher score means a worse outcome.
Psychological resilience | 12 months, 24 months and 36 months
  Measure by the 10-Items Connor-Davidson Resilience Scale (CD-RISC-10), scoring from 0-40 and a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, The Chinese University of Hong Kong (CUHK), Ward 3M, Diabetes and Endocrine Research Centre, 3/F Day Treatment Block and Children Wards (Old Block), Prince of Wales Hospital, Hong Kong, Hong Kong